CLINICAL TRIAL: NCT04440345
Title: Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IBI362 in Overweight or Obese Subjects
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IBI362 in Overweight or Obesity Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362B101
Record Dates: First submitted 2020-06-05; First posted 2020-06-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI362 (Experimental): Participants received dose 1 level of IBI362 administered as multiple subcutaneous doses.
  Participants received dose 2 level of IBI362 administered as multiple subcutaneous doses.
  Participants received dose 3 level of IBI362 administered as multiple subcutaneous doses.
  Participants received dose 4 level of IBI362 administered as multiple subcutaneous doses.
  Participants received dose 5 level of IBI362 administered as multiple subcutaneous doses.
  Interventions: Drug: IBI362
- placebo (Placebo Comparator): Participants received matching placebo dose regiments by subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBI362 — Administered by subcutaneous injection
  Arms: IBI362
Drug: Placebo — Administered by subcutaneous injection
  Arms: placebo

SUMMARY:
This trial is conducted in China. The aim of this trial is to investigate Safety, Tolerability, PK and PD for Multiple Doses of IBI362 in Overweight or Obese Male and Female Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have stable body weight for the past 12 weeks prior to screening
2. Have a body mass index (BMI) ≥24 kilograms per meter squared (kg/m²) with complication, or BMI≥28 kg/m²,inclusive at screening
3. Willing and agreeable to commit to the duration of the study and undergo study procedures as instructed by the clinic staff

Exclusion Criteria:

1. Have a diagnosis of type 2 diabetes
2. Have received prescription drugs or over the counter drugs that promote weight loss in the past 3 months prior to screening
3. Previous treatment with a GLP-1 (glucagon-like peptide 1) receptor agonists or GCG(glucagon)receptor agonists before.
4. Surgical treatment for obesity
5. Past or current chronic or idiopathic pancreatitis, or any of the following: -amylase or lipase above 2 times UNR (upper normal range), triglycerides above 500 mg/dL
6. Have other medical conditions or medical history that make participation in the study unsafe or which may interfere in the interpretation of the results of the study
7. Unwilling to comply with smoking and alcohol restrictions during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Number of treatment adverse events | From the time of first dosing (Day 1 ) until completion of the post treatment follow-up visit (20 week)
  The relationship of each adverse event to the investigational product was assessed by the investigator.

SECONDARY OUTCOMES:
Number of Participants With Anti-IBI362 Antibodies | From the time of first dosing (Day 1 )until comletion of the post treatment follow-up visit (20 week)
  Serum samples were analyzed by an electrochemiluminescence (ECL)-based immunoassay for anti-IBI362 binding antibodies. Positive samples were subsequently tested in a receptor-ligand binding bioassay for anti-IBI362 neutralizing antibodies.
Evaluate the Peak Plasma Concentration (Cmax) of IBI362 in overweight or obesity subjects; | From the first dose (Day 1 ) of study drug until 12 week
Evaluate the Area under the plasma concentration versus time curve (AUC) of IBI362 in overweight or obesity subjects; | From the first dose (Day 1 ) of study drug until 12 week
Evaluate the Fasting Blood Glucose (FBG ) of IBI362 in overweight or obesity subjects; | From the first dose (Day 1 ) of study drug until 12 week
Evaluate the Glucagon of IBI362 in overweight or obesity subjects; | From the first dose (Day 1 ) of study drug until 12 week
Evaluate the Insulin of IBI362 in overweight or obesity subjects; | From the first dose (Day 1 ) of study drug until 12 week
Evaluate the C-peptide of IBI362 in overweight or obesity subjects; | From the first dose (Day 1 ) of study drug until 12 week
Change in body weight from baseline | Baseline (Day 1 ) and 12 week for groups

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University people's hospital, Beijing, China

REFERENCES:
- [Derived] Ji L, Gao L, Jiang H, Yang J, Yu L, Wen J, Cai C, Deng H, Feng L, Song B, Ma Q, Qian L. Safety and efficacy of a GLP-1 and glucagon receptor dual agonist mazdutide (IBI362) 9 mg and 10 mg in Chinese adults with overweight or obesity: A randomised, placebo-controlled, multiple-ascending-dose phase 1b trial. EClinicalMedicine. 2022 Oct 7;54:101691. doi: 10.1016/j.eclinm.2022.101691. eCollection 2022 Dec. PMID 36247927
- [Derived] Ji L, Jiang H, An P, Deng H, Liu M, Li L, Feng L, Song B, Han-Zhang H, Ma Q, Qian L. IBI362 (LY3305677), a weekly-dose GLP-1 and glucagon receptor dual agonist, in Chinese adults with overweight or obesity: A randomised, placebo-controlled, multiple ascending dose phase 1b study. EClinicalMedicine. 2021 Aug 13;39:101088. doi: 10.1016/j.eclinm.2021.101088. eCollection 2021 Sep. PMID 34430840